CLINICAL TRIAL: NCT04555252
Title: Colonization of Bile Ducts and Post-operative Infectious Complications of Cephalic Duodenopancreatectomy : A Prospective Observational Study
Brief Title: Colonization of Bile Ducts and Infectious Complications in Cephalic Duodenopancreatectomy
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: CHRU NANCY : 2019PI249
Record Dates: First submitted 2020-08-10; First posted 2020-09-18 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2020-07

CONDITIONS: Infection, Bacterial
Keywords: Bile colonization; Cephalic Duodenopancreatectomy
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cephalic Duodenopancreatectomy: Patients who underwent scheduled cephalic duodenopancreatectomy and hospitalized in intensive care.

SUMMARY:
Cephalic duodenopancreatectomy is part of the curative treatment for pancreatic cancer of the head and peri-ampullary area. The mortality of the procedure is around 5%, with a morbidity ranging from 30 to 50%. Infectious complications account for 35% of overall morbidity.

One of the risk factors for postoperative complications is the existence of preoperative retentional jaundice, due to tumoral obstruction of the main bile duct In these cases, it is proposed to perform preoperative bile duct drainage, preferably by endoscopic stenting (ERCP).

However, several studies have shown these procedures to cause biliary contamination which could be responsible for an increase in post-operative morbidity such as infectious complications and increased length of stay in hospital..

Thus, the biliary microbial flora is more often multi-microbial and may contain multidrug-resistant nosocomial germs,

The study carried out by Cortes et al., based on a control case study design, also showed that a correlation between biliary colonization and postoperative infectious complications existed in patients who benefited from a preoperative biliary drainage technique. In fact, the bacteria isolated during intraoperative bile sampling were similar, in 49% of cases, to those isolated during bacteriological samples collected postoperatively during infectious complications.

The work carried out by Krüger and al has shown that the spectrum of bacteria found in the preoperative bile samples from patients who have undergone bile duct dilation is potentially not covered by standard antibiotic therapy.

The aim of this observational prospective study is to investigate this correlation between biliary colonization and postoperative infectious complications, to evaluate the morbidity and postoperative mortality of cephalic duodenopancreatectomies performed at the CHRU of Nancy and to study a possible adaptation of perioperative antibiotic prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient operated for a planned cephalic duodenopancreatectomy
* Post-operative hospitalisation in ICU
* Information leaflet given to the patient and the support person, with oral information, during the post-operative period

Exclusion Criteria:

* Age < 18 years
* Emergency duodenopancreatectomy (surgical indication period less than 48 hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be offered to the patient who has benefited from a cephalic duodenopancreatectomy programmed and hospitalized in CHRU Nancy's ICU
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-03-28 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Comparison of preoperative Bile and postoperative infection sites microbiology results | from date of initial bile sample up to 30 days of postoperative period
  bacterial count in log10 bacteria/ml and identification

SECONDARY OUTCOMES:
Impact of prior biliary drainage on the intraoperative bile microbiological results bacteriological results obtained | from date of initial bile sampling to date of surgery (up to 90 days)
  bacterial count in log10 bacteria/ml and species identification
Microbial flora in clinical specimens obtained from different sites | from date of initial bile sample up to 90 postoperative days
  bacterial count in log10 bacteria/ml and species identification
Non infectious surgical complications using scores | from date of surgery up to 30 postoperative days
  Clavien-Dindo Classification, SOFA score
postoperative infectious complications as defined by the Centers for Disease Control and Prevention (Atlanta, Ga) | During hospital stay (up to 90 days after surgery)
  number of event occurence
Implication of bacteria found in biliculture as causative agent in post-operative infections | During hospital stay (up to 90 days after surg
  incidence in percentage
length of stay in intensive care and hospital | During the ICU stay and hospital
  Number of days in ICU and hospital
mortality rate | At day +28 and day +90
  number of death at 28 days and 90 days
Description of nutrition assistance | from date of initial bile sample up to 30 days of postoperative period
  Parenteral, enteral, oral feeding in days and calories
Nutritional status measured by nutritional risk index (NRI) | preoperative
  Body mass index (BMI) and albuminemia computation

CONTACTS AND LOCATIONS:
Overall Officials: MARIE-REINE LOSSER, MD,PhD, Principal Investigator — CHRU Nancy
Locations (1):
- Chru Nancy, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Background] Ho V, Heslin MJ. Effect of hospital volume and experience on in-hospital mortality for pancreaticoduodenectomy. Ann Surg. 2003 Apr;237(4):509-14. doi: 10.1097/01.SLA.0000059981.13160.97. PMID 12677147
- [Background] DeOliveira ML, Winter JM, Schafer M, Cunningham SC, Cameron JL, Yeo CJ, Clavien PA. Assessment of complications after pancreatic surgery: A novel grading system applied to 633 patients undergoing pancreaticoduodenectomy. Ann Surg. 2006 Dec;244(6):931-7; discussion 937-9. doi: 10.1097/01.sla.0000246856.03918.9a. PMID 17122618
- [Background] Okano K, Hirao T, Unno M, Fujii T, Yoshitomi H, Suzuki S, Satoi S, Takahashi S, Kainuma O, Suzuki Y. Postoperative infectious complications after pancreatic resection. Br J Surg. 2015 Nov;102(12):1551-60. doi: 10.1002/bjs.9919. Epub 2015 Sep 21. PMID 26387569
- [Background] Yu L, Huang Q, Xie F, Lin X, Liu C. Risk factors of postoperative complications of pancreatoduodenectomy. Hepatogastroenterology. 2014 Oct;61(135):2091-5. PMID 25713915
- [Background] Lermite E, Pessaux P, Teyssedou C, Etienne S, Brehant O, Arnaud JP. Effect of preoperative endoscopic biliary drainage on infectious morbidity after pancreatoduodenectomy: a case-control study. Am J Surg. 2008 Apr;195(4):442-6. doi: 10.1016/j.amjsurg.2007.03.016. PMID 18304506
- [Background] Scheufele F, Aichinger L, Jager C, Demir IE, Schorn S, Sargut M, Erkan M, Kleeff J, Friess H, Ceyhan GO. Effect of preoperative biliary drainage on bacterial flora in bile of patients with periampullary cancer. Br J Surg. 2017 Jan;104(2):e182-e188. doi: 10.1002/bjs.10450. PMID 28121036
- [Background] Cortes A, Sauvanet A, Bert F, Janny S, Sockeel P, Kianmanesh R, Ponsot P, Ruszniewski P, Belghiti J. Effect of bile contamination on immediate outcomes after pancreaticoduodenectomy for tumor. J Am Coll Surg. 2006 Jan;202(1):93-9. doi: 10.1016/j.jamcollsurg.2005.09.006. Epub 2005 Nov 18. PMID 16377502
- [Background] Kruger CM, Adam U, Adam T, Kramer A, Heidecke CD, Makowiec F, Riediger H. Bacterobilia in pancreatic surgery-conclusions for perioperative antibiotic prophylaxis. World J Gastroenterol. 2019 Nov 7;25(41):6238-6247. doi: 10.3748/wjg.v25.i41.6238. PMID 31749594